CLINICAL TRIAL: NCT07131020
Title: Study on the Mechanism of Yifei Moxibustion in Enhancing Immune Function in Chronic Obstructive Pulmonary Disease Based on Plasma Exosomal miRNAs
Brief Title: Study on the Mechanism of Yifei Moxibustion Improving Immune Function in COPD Based on Plasma Exosome miRNAs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yifei moxibustion for COPD
Record Dates: First submitted 2025-08-10; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Stable COPD Patients
Keywords: COPD; Yifei moxibustion; miR-125b; macrophage polarization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yifei moxibustion group (Experimental): The patients in the Yifei Moxibustion group are treated with conventional Western medicine combined with Yifei Moxibustion.
  Interventions: Behavioral: Yifei moxibustion
- Conventional Western medicine treatment group (Active Comparator): The patients in the conventional Western medicine treatment group receives standard Western medication therapy.
  Interventions: Drug: Conventional Western medicine treatment
- TCM syndrome differentiation treatment group (Active Comparator): Patients in the TCM syndrome differentiation treatment group receives TCM pattern-based therapy in addition to conventional Western medical treatment.
  Interventions: Drug: TCM syndrome differentiation treatment

INTERVENTIONS:
Behavioral: Yifei moxibustion — The conventional Western medicine treatment is based on the 2023 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and the 2021 Chinese Thoracic Society guidelines for the diagnosis and management of chronic obstructive pulmonary disease. Bronchodilators, inhaled corticosteroids, or a combination therapy are administered.The Yifei moxibustion is applied from the Dazhui to Yaoshu acupoints along the Governor Vessel. Ginger juice is spread over the treatment area, followed by sprinkling moxa powder and covering with mulberry bark paper. A 2.5 cm thick layer of ginger paste and a 3 cm thick layer of moxa wool are then placed on the mulberry bark paper. The moxa wool is ignited and allowed to burn out naturally, being replaced every 30 minutes. After 90 minutes, the ginger paste is removed. The treatment is performed once every 15 days, with 6 sessions constituting one course of treatment, totaling 3 months.
  Arms: Yifei moxibustion group
Drug: Conventional Western medicine treatment — The conventional Western medicine treatment is based on the 2023 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and the 2021 Chinese Thoracic Society guidelines for the diagnosis and management of chronic obstructive pulmonary disease. Bronchodilators, inhaled corticosteroids, or a combination therapy are administered.
  Arms: Conventional Western medicine treatment group
Drug: TCM syndrome differentiation treatment — The conventional Western medicine treatment followes the same protocol as described above. The diagnosis of TCM pattern-based therapy is made in accordance with the TCM Syndrome Diagnostic Criteria for Chronic Obstructive Pulmonary Disease issued by the Pulmonary Disease Committee of the Internal Medicine Branch, China Association of Chinese Medicine and the treatment is based on the 2019 Guidelines for Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease issued by the China Association of Chinese Medicine.
  Arms: TCM syndrome differentiation treatment group

SUMMARY:
This study adopted a randomized controlled design, enrolling 90 patients and 30 healthy volunteers. The patients were randomly divided into the Yifei Moxibustion group, the conventional Western medicine treatment group, and the TCM syndrome differentiation treatment group, and were treated for 3 months. Peripheral venous blood was collected from both the healthy volunteers and the patients to observe indicators such as T cell subsets and immunoglobulins, to evaluate the effect of Yifei Moxibustion on improving immune function. The regulation of target genes by exosomes and potential action targets and molecular mechanisms were preliminarily verified through techniques such as nanoparticle tracking technology and flow cytometry.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the most common chronic airway disease, and airway inflammation and immune regulation mechanisms play a significant role in its development. Macrophage polarization is involved in the immune response process of COPD and is crucial for the resolution of airway inflammation and the regulation of the body's immune system. Among them, M1 polarization of macrophages can expand the inflammatory response, cause tissue damage, and aggravate the disease progression. Literature indicates that exosomal miR-125b may be an important target for regulating M1 polarization of macrophages.Yifei Moxibustion can improve the immune function of COPD patients, but its mechanism of action is still unclear. Therefore, the following hypothesis is proposed: Yifei Moxibustion can promote the resolution of inflammation and regulate the body's immune system by regulating miR-125b-mediated M1 polarization of macrophages. This study adopts a randomized controlled design, including 90 patients and 30 healthy volunteers. Patients are randomly divided into the Yifei Moxibustion group, the Western medicine conventional treatment group, and the TCM syndrome differentiation treatment group, and treated for 3 months. Peripheral venous blood is collected from healthy volunteers and patients. Firstly, T cell subsets, immunoglobulins and other indicators are observed to evaluate the effect of Yifei Moxibustion on improving immune function. Secondly, macrophage polarization is detected by nanoparticle tracking analysis, co-culture of transfected cells, CCK8 and other methods. miR-125b differentially expressed target genes are screened by miRDB and other databases, and the secretion of target genes regulated by exosomes is verified by luciferase reporter gene and other methods. Finally, macrophage polarization-related markers of patients before and after intervention are detected by flow cytometry, ELISA and other methods to preliminarily verify the regulation of exosomes on target genes, as well as potential targets and molecular mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for stable chronic obstructive pulmonary disease;

  * Patients who meet the TCM diagnostic criteria for lung qi deficiency, lung-spleen qi deficiency, and lung-kidney qi deficiency; ③ Aged 18 to 80 years old; ④ Voluntarily signed the informed consent form.

Exclusion Criteria:

* Pregnant and lactating women;

  * Patients with cognitive impairment, confusion, dementia, or various mental disorders;

    * Patients with unstable angina pectoris or acute myocardial infarction;

      * Patients with a history of syncope after exercise or bone and joint diseases that affect exercise; ⑤ Patients with pneumothorax, pleural effusion, pulmonary embolism, or tumors;

        * Patients known to be allergic to the ingredients of the moxibustion powder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The level of plasma exosomal miR-125b | Before treatment and 3 months after treatment
  The regulatory effect of Yifei moxibustion on miR-125b was evaluated through the detection of peripheral venous blood.
T-cell subsets and immunoglobulin levels | Before treatment and 3 months after treatment
  By detectingCD3+、CD4+、CD8+、CD4+/CD8+、Th17、Treg、Th17/Treg 、IgG、IgA、IgM, the regulatory effect of Yifei moxibustion on the immune function of COPD was evaluated.

SECONDARY OUTCOMES:
Clinical Symptoms and Signs Assessment Questionnaire Assessment | Before treatment, the first month, the second month and the third month
  Clinical Symptoms and Signs Assessment Questionnaire Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, phlegm, chest tightness, gasp, shortness of breath, feeble and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
The modified Medical Research Council (mMRC) scale | Before treatment, the first month, the second month and the third month
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
lung function | Time Frame：Before treatment and 3 months after treatment
  Forced Vital Capacity (FVC)#Forced Expiratory Volume in One Second (FEV1) and Percentage of Forced Expiratory Volume in One Second to Predicted Value (FEV1% pred) were mainly used for lung function evaluation
Six-Minute Walk Distance（6MWD） | Before treatment, the first month, the second month and the third month
  The six-minute walk distance is used to assess exercise tolerance and functional status.
The COPD Assessment Test (CAT) | Before treatment, the first month, the second month and the third month
  The COPD Assessment Test (CAT) is an 8-item questionnaire that assesses health status in patients with COPD. The questionnaire uses a 0-5 point scale, with higher values indicating a greater impact of COPD on the patient.
The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) | Before treatment, the first month, the second month and the third month.
  The modified COPD Patient-Reported Outcome scale (mCOPD-PRO) will be used to assess quality of life. The mCOPD-PRO contains 27 items in three domains. mCOPD-PRO scores range from 0 to 4 with a decrease in score showing higher health status.
The modified Effectiveness Satisfaction Questionnaire for COPD | Before treatment, the first month, the second month and the third month
  (mESQ-COPD)The modified Effectiveness Satisfaction Questionnaire for COPD (mESQ-COPD) will be used to assess treatment satisfaction. The mESQ-COPD contains 19 items in four domains. mESQ-COPD scores range from 0 to 4 with a decrease in score showing higher treatment satisfaction.
Acute exacerbation situation | Before treatment, the first month, the second month and the third month
  The frequency of colds and acute exacerbations was used to assess the improvement of immune function in patients with chronic obstructive pulmonary disease by Yifei moxibustion.
Adverse Event Documentation and Laboratory Safety Metrics | Before treatment and 3 months after treatment
  Adverse Event Documentation and aboratory safety indicators such as blood routine, urine routine, liver function, kidney function, electrocardiogram are used to assess the safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xie, Doctor, Principal Investigator — the First Affiliated Hospital of Henan University of Chinese Medicine
Locations (1):
- the First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No